CLINICAL TRIAL: NCT06051877
Title: Ocular Microtremor in Parkinson's Disease
Acronym: OMTinPD
Status: Recruiting | Type: Observational
Sponsor: Northumbria University (Other)
Collaborators: Northumbria Healthcare NHS Foundation Trust (Other); Gateshead Health NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: OMT in PD
Record Dates: First submitted 2023-09-18; First posted 2023-09-25 (Actual); Last update posted 2024-04-19 (Actual); Status verified 2024-04

CONDITIONS: Parkinson's Disease; Parkinson Disease
Keywords: Ocular microtremor; Eye movements; Biomarker; Parkinson's Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Week
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- suspPD: People referred to clinic with suspected PD
- confPD: People with confirmed PD
- HC: Healthy controls

SUMMARY:
This is an exploratory, observational study that will use a novel handheld device - The iTremor ONE, which has been developed to rapidly, non-invasively assess and evaluate OMT frequency. This device uses incident laser technology directed at the sclera. PwPD who meet the inclusion criteria will participate in a home-based assessment involving cognitive, motor (using the UPDRS-III) and OMT measures. With OMT as the primary outcome, assessment with the iTremor is incredibly quick, taking just three seconds to obtain a reading. PwPD will be assessed both 'off' and on their anti-parkinsonian medication. 'Off' is defined as a 12Hr overnight washout period where participants are tested in the morning prior to their first dose. PwPD will also be invited into the laboratory to perform extensive cognitive assessments along with an assessment of balance, gait, and turning using wearable sensors. 40 PwPD, 20 with suspected PD, and 40 age-matched healthy control participants will be recruited for assessment of OMT. Ten PwPD will complete a test-retest reliability assessment at the same approx. time, exactly one week after their initial visit.

DETAILED DESCRIPTION:
Ocular microtremor (OMT) is a fixational eye movement that cannot be seen with the naked eye but is always present, even when the eye appears motionless/still. The link between OMT and brain function generates a strong rationale for investigation as there lies potential for its use as a biomarker in populations of neurological impairments. OMT frequency is typically 70-80Hz in healthy adults and research suggests that this will be reduced in those with neurological disease such as Parkinson's Disease (PD). This study aims to examine OMT in people with PD (PwPD) compared to healthy older adults. Identifying OMT as a PD biomarker could better support clinical assessment, enabling improved provision of care to patients with advanced disease monitoring.

This is an exploratory, observational study that will use a novel handheld device - The iTremor ONE, which has been developed to rapidly, non-invasively assess and evaluate OMT frequency. This device uses incident laser technology directed at the sclera. PwPD who meet the inclusion criteria will participate in a home-based assessment involving cognitive, motor (using the UPDRS-III) and OMT measures. With OMT as the primary outcome, assessment with the iTremor is incredibly quick, taking just three seconds to obtain a reading. PwPD will be assessed both off and on their anti-parkinsonian medication. PwPD will also be invited into the laboratory to perform extensive cognitive assessments along with an assessment of balance, gait, and turning using wearable sensors. The Investigators will recruit 40 PwPD, 20 suspected PD, and 30 age-matched healthy control participants for assessment of OMT. Ten PwPD will complete a test-retest reliability assessment at the same approx. time, exactly one week after their initial visit.

This will be the first study of its kind to non-invasively investigate OMT frequency as a marker/monitor for PD with advanced technology that could be used within the clinic, laboratory, or home.

ELIGIBILITY:
Inclusion Criteria:

* People with suspected PD
* People with confirmed PD
* Healthy controls
* No history of head trauma

Exclusion Criteria:

* PD and older adult participants will be excluded if there is any psychiatric co-morbidity,
* a history or evidence of head injury or ocular disease (such as cataracts),
* they have a clinical diagnosis of dementia or other severe cognitive impairment (measured using the MoCA with a score of <21).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants will be a volunteer sample recruited from Northumbria Healthcare and Gateshead Health NHS foundation trusts. These clinics are run by Professor Richard Walker and Dr Claire McDonald (consultant geriatricians) respectively. Participants will be seen in clinic by a Movements Disorders specialist at these sites where people referred for suspected PD diagnosis and those with diagnosed PD will be identified. Potential participants will be invited to consider the study and referred to the investigators who will attend the clinics. Healthy controls could include spouses/ siblings/ other volunteer older adults.
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2024-09-30 (Estimated); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
OMT frequency (Hz) | 2 weeksw
  Ocular mictoremor frequency (Hz) as measures with the iTremor ONE device

CONTACTS AND LOCATIONS:
Overall Officials: Samuel Stuart, PhD, Principal Investigator — Employee
Locations (2):
- United Kingdom (2):
  - Gateshead Health NHS Foundation Trust, Gateshead, Tyne and Wear
  - Northumbria Healthcare NHS Trust, North Shields, Tyne and Wear

IPD SHARING:
Plan to Share IPD: No
There is no plan to make IPD available.

REFERENCES:
- [Derived] Graham L, Vitorio R, Walker R, Godfrey A, Morris R, Stuart S. Digital measurement of ocular microtremor in Parkinson's disease: Protocol for a pilot study to assess reliability and clinical validation. PLoS One. 2025 Jan 8;20(1):e0313452. doi: 10.1371/journal.pone.0313452. eCollection 2025. PMID 39775540